CLINICAL TRIAL: NCT05243797
Title: Phase 3 Study of Teclistamab in Combination With Lenalidomide and Teclistamab Alone Versus Lenalidomide Alone in Participants With Newly Diagnosed Multiple Myeloma as Maintenance Therapy Following Autologous Stem Cell Transplantation - MajesTEC-4
Brief Title: Phase 3 Study of Teclistamab in Combination With Lenalidomide and Teclistamab Alone Versus Lenalidomide Alone in Participants With Newly Diagnosed Multiple Myeloma as Maintenance Therapy Following Autologous Stem Cell Transplantation
Acronym: MajesTEC-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN30/64007957MMY3003
Record Dates: First submitted 2022-01-27; First posted 2022-02-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Maintenance; Teclistamab
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: Teclistamab-Lenalidomide (Tec-Len) (Experimental): Teclistamab will be administered via a subcutaneous injection (SC)
  Interventions: Drug: Teclistamab; Drug: Lenalidomide
- Arm B Lenalidomide Alone (Len) (Active Comparator): Lenalidomide orally.
  Interventions: Drug: Lenalidomide
- Arm C Teclistamab-Alone (Tec) (Experimental): Teclistamab will be administered via a subcutaneous injection (SC)
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered via a subcutaneous injection (SC)
  Other Names: JNJ-64007957
  Arms: Arm A: Teclistamab-Lenalidomide (Tec-Len); Arm C Teclistamab-Alone (Tec)
Drug: Lenalidomide — Lenalidomide will be administered orally
  Arms: Arm A: Teclistamab-Lenalidomide (Tec-Len); Arm B Lenalidomide Alone (Len)

SUMMARY:
This is a multicenter, randomized, open-label, Phase 3 study in participants with newly diagnosed multiple myeloma to evaluate the benefits of teclistamab in combination with lenalidomide and teclistamab alone versus lenalidomide alone as maintenance therapy after autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Must have a new diagnosis of multiple myeloma according to IMWG criteria and have received induction +/- consolidation.
* Must have received only one line of therapy and achieved at least a partial response (≥PR) as per IMWG 2016 response criteria (Kumar 2016) without evidence of progression at the time of first treatment dose.
* Must not be intolerant to the starting dose of lenalidomide.
* Must not have received any maintenance therapy.
* Have an ECOG performance status score of 0, 1, or 2 at screening and immediately prior to the start of administration of study treatment
* Have clinical laboratory values within prespecified range.

Exclusion Criteria:

* Received any prior BCMA-directed therapy.
* Any previous therapy with an immune cell redirecting agent or gene modified adoptive cell therapy (eg, chimeric antigen receptor modified T cells, NK cells).
* Discontinued treatment due to any AE related to lenalidomide as determined by the investigator.
* Progressed on multiple myeloma therapy at any time prior to screening.
* Received a cumulative dose of corticosteroids equivalent to ≥140 mg of prednisone within the 14 days prior to first treatment dose.
* Received a live, attenuated vaccine within 4 weeks before first treatment dose. Non-live vaccines or non-replicating authorized for emergency use (eg. COVID-19) are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1594 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | from randomization to the date of disease progression or death (approximately up to 8 years)
  PFS is defined as the time from the date of randomization to the date of disease progression (as assessed by IMWG criteria) or death due to any cause, whichever occurs first.
Minimal Residual Disease (MRD)-negative Complete Response (CR) | at month 12
  12-month MRD-negative CR is defined as participants who achieve MRD-negative status at 12 months, as determined by next-generation flow cytometry (NGF) with sensitivity of 10^-5, prior to progressive disease or subsequent anti-myeloma therapy, whichever is earlier, and who also achieve CR of better, according to IMWG criteria.

SECONDARY OUTCOMES:
Comparison of efficacy | from randomization to the date of disease progression or death (approximately up to 8 years)
  Efficacy, assessed by rate of CR or better, MRD negative CR, sustained MRD negativity, CR and MRD negative conversion PFS after next line of therapy (PFS2), time to next treatment (TTNT), OS and also safety, PK and immunogenicity
Overall Survival (OS) | from the date of from randomization to the date the subject's death, assessed up to 8 years]
  Overall Survival (OS), measured from the date of from randomization to the date the subject's death
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core module (EORTC QLQ-C30) score and the difference between-treatment arms | baseline up to 8 years
  The EORTC QLQ-C30 is a 30-item questionnaire containing both single and multi-item measures. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/ Quality-of-Life (QoL) scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). The scores ranges from 0-100, a high score for functional scales and for Global Health Status/QoL represent better functioning ability or Health-Related Quality-of-Life (HRQoL), whereas a high score for symptom scales and single items represents significant symptomatology.
EQ-5D-5L health utility values and the difference between-treatment arms | baseline up to 8 years
  The EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today"
MySIm-Q Symptom and Impacts in Patients With Multiple Myeloma and the difference between treatment arms | baseline up to 8 years
  The MySIm-Q is a disease-specific PRO assessment complementary to the EORTC-QLQ-C30. It includes 17 items resulting in a symptom subscale and an impact subscale. The recall period is the "past 7 days", and responses are reported on a 5-point verbal rating scale.
PRO-CTCAE to evaluate symptomatic toxicities by self-report and the difference between treatment arms | baseline up to week 24
  The PRO-CTCAE Measurement System characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities. The PRO-CTCAE Item Library includes 124 items representing 78 symptomatic toxicities drawn from the CTCAE
PGIS to evaluate the patient global impression of severity of the Multiple Myeloma and the difference between treatment arms | baseline up to 8 years
  PGIS is a 1 item questionnaire that evaluates patients' health and assesses if there has been an improvement or decline in clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Niels van de Donk, Professor, Principal Investigator — Amsterdam UMC, Vrije Universiteit Amsterdam; Elena Zamagni, Professor, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna, Istituto di Ematologia "Seràgnoli"
Locations (208):
- United States (38):
  - Banner University Medical Center Tucson, University of Arizona, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - University of California-Davis Cancer Center, Sacramento, California
  - University of California, San Diego (UCSD) Medical Center, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Care, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Blood & Marrow Transplant Center, Florida Hospital Medical Group, Orlando, Florida
  - Moffitt at Memorial Healthcare System, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Illinois Medical Center at Chicago, Chicago, Illinois
  - Greenebaum Cancer Center UM of MD, Baltimore, Maryland
  - John Hopkins, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Mount Sinai Medical Center - 2, New York, New York
  - Montefiore Medical Cente, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Seidman Cancer Center-University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State Medical Center, James Cancer Center, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Abramson Cancer Center University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Vanderbilt-Ingram Cancer Center (VICC), Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - St Vincent HSHS (Green Bay Oncology), Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Italiano, Buenos Aires
  - Hospital Privado, Córdoba
  - Sanatorio Britanico Rosario, Rosario
- Australia (10):
  - Sunshine Coast Health, Birtinya, Queensland
  - Flinders Medical Centre, Adelaide
  - Townsville University Hospital, Douglas
  - Barwon Health University Hospital Geelong Andrew Love Cancer Centre, Geelong
  - Alfred Hospital, Melbourne
  - Austin Health, Melbourne
  - Calvary Mater Hospital, Newcastle
  - Sunshine Coast Health, Sunshine Coast
  - Concord Repatriation General Hospital, Sydney
  - Royal North Shore Hospital, Sydney
- Austria (8):
  - Landeskrankenhaus, Feldkirch, Feldkirch
  - Medizinische Universitaet Innsbruck, Innsbruck
  - University Hospital Krems/Donau, Krems
  - Kepler Universitätsklinikum Med Campus III, Linz
  - Ordensklinikum Linz GmbH, Linz
  - Uniklinikum Salzburg, Salzburg
  - Clinic Ottakring, Vienna
  - LKH Hochsteiermark, Vienna
- Belgium (5):
  - Jessa Ziekenhuis, Hasselt
  - Department of Hematology, CH Jolimont, La Louvière
  - Algemeen Ziekenhuis Delta, Leuven
  - University Hospital Leuven, Leuven
  - Centre hospitalier universitaire de Liege, Liège
- Brazil (14):
  - Hospital Mãe de Deus - Centro Integrado de Oncologia, Porto Alegre
  - Hospital Santa Rita, Porto Alegre
  - Instituto Americas de Ensino,Pesquisa e Inovação, Rio de Janeiro
  - IDOR- Instituto D'or de pesquisa. Av. São Rafael, Salvador
  - A Real e Benemérita Associação Portuguesa de Beneficência, São Paulo
  - Clínica Medica São Germano,Grupo Oncoclínicas Pesquisa Clínica, São Paulo
  - Departamento de Oncologia Clínica AC Camargo Cancer Center, São Paulo
  - Grupo Oncoclínicas Pesquisa Clínica, São Paulo
  - Hcor, Associacao Siria, São Paulo
  - Hemocentro UNICAMP, Universidade Estadual de Campinas, São Paulo
  - Hospital das Clínicas da Universidade de São Paulo, São Paulo
  - Hospital Paulistano, Centro de Pesquisa Clinica R. Martiniano de Carvalho, São Paulo
  - Onco Star, São Paulo
  - Universidade Federal de São Paulo - Hospital São Paulo, São Paulo
- Canada (7):
  - Cross Cancer Institute, Edmonton
  - QEII Health Sciences Centre, Halifax
  - The Ottawa General Hospital, Ottawa
  - Saskatoon Cancer Center, Saskatoon
  - "Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke (CIUSSS de l'Estrie - CHUS)", Sherbrooke
  - Princess Margaret Cancer Centre, Toronto
  - BC Cancer, Vancouver
- China (11):
  - Beijing Chaoyang Hospital, Beijing
  - Peking University First Hospital, Beijing
  - North China University of Science and Technology Affiliated Hospital.Hematology Department, Hebei
  - Henan Cancer Hospital, Henan
  - Shandong Qilu Hospital, Shandong
  - Shanghai Fourth People's Hospital, Shanghai
  - Shenyang City, Liaoning Province, Hematology department, Shenyang
  - Institute of Hematology & Blood Disease Hospital Chinese Academy of Medical Science, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital, Tongji Medical College of Hust, Wuhan
  - The First Affiliated Hospital, Zhejiang University College of Medicine, Zhejiang
- Czechia (5):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni Nemocnice Plzen, Pilsen
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- Denmark (4):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Lillebaelt Hospital, Vejle
- France (9):
  - Centre Hospitalier Universitaire De Bordeaux, Bordeaux
  - Department of Hematology, CHU Lille, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Universitaire De Montpellier, Montpellier
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Hopital Saint Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Centre Hospitalier Universitaire De Poitiers, Poitiers
  - Centre Hospitalier Universitaire De Toulouse, Toulouse
- Germany (8):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg AöR, Heidelberg
  - Universitaetsklinikum Jena KöR, Jena
  - Universitaetsklinikum Schleswig-Holstein AöR, Lübeck
  - Klinikum rechts der Isar der TU Muenchen AöR, München
  - Klinikum Nuernberg, Nuremberg
  - Universitaetsklinikum Tuebingen AöR, Tübingen
  - University Hospital of Würzburg, Würzburg
- Greece (4):
  - University General Hospital Of Alexandroupoli, Alexandroupoli
  - Evaggelismos Hospital, Athens
  - Regional General Hospital Alexandra, Athens
  - Theageneio Cancer Hospital, Thessaloniki
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
- Israel (6):
  - The Barzilai Medical Center, Beersheba
  - Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Beilinson Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (28):
  - Azienda Sanitaria Locale Al Di Alessandria, Alessandria
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I G M Lancisi G Salesi, Ancona
  - AOU G. Baccelli, Bari
  - Policlinico di Bari, Bari
  - A.O. Papa Giovanni XXIII, Bergamo
  - A.O.U. di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - A.O.Spedali Civili di Brescia, Brescia
  - Ospedale Oncologico 'A. Businco', Cagliari
  - Azienda Ospedaliera-Universitaria Di Cosenza, Cosenza
  - Careggi University Hospital, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova
  - IRCCS Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero Universitaria Di Modena, Modena
  - Azienda Ospedaliera Di Rilievo Nazionale Antonio Cardarelli, Napoli
  - UOC Oncoematologia, Ospedale Policlinico Federico II, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore Della Carita, Novara
  - UOC Ematologia - Azienda Ospedale - Università Padova Ospedale Giustinianeo, Padua
  - Department of Hematology and Bone Marrow Transplant Centre, Azienda Ospedaliero - Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Sanitaria Locale Di Pescara, Pescara
  - Ospedale Santa Maria delle Croci, Ravenna
  - Azienda USL IRCCS Di Reggio Emilia, Reggio
  - Ospedale "Infermi" di Rimini, Rimini
  - Ematologia, Azienda Policlinico Umberto I, Roma
  - Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - A.O.U. Città della Salute e della Scienza di Torino - SC Ematologia U, Torino
  - A.O.U. Ospedali Riuniti di Trieste, Trieste
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Netherlands (9):
  - Noordwest Ziekenhuisgroep Stichting, Alkmaar
  - Amsterdam University Medical Center, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Maxima Medisch Centrum, Eindhoven
  - University Medical Center Groningen, Groningen
  - Dijklander Ziekenhuis, Hoorn
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus University Medical Center Rotterdam, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
- St. Olavs hospital HF, Trondheim, Norway
- Poland (2):
  - Department of Hematology and Transplantology University Clinical Center, Gdansk
  - SPZOZ MSWiA w Poznaniu im. Prof. Ludwika Bierkowskiego, Poznań, Poznan
- Portugal (7):
  - CCAB Centro Clinico Academico Braga Associacao, Braga
  - Champalimaud Clinical Centre, Lisbon
  - Instituto Portugues De Oncologia De Lisboa Francisco Gentil E.P.E., Lisbon
  - Instituto Portugues De Oncologia Do Porto Francisco Gentil E.P.E., Porto
  - Sao Joao University Hospital Center, Porto
  - Unidade Local De Saude De Gaia/Espinho E.P.E., Porto
  - Unidade Local De Saude De Tras-Os-Montes E Alto Douro E.P.E., Vila Real
- Serbia (4):
  - University Clinical Center of Serbia, Belgrade
  - Clinical Centre of Kragujevac, Kragujevac
  - Clinical Centre of Nis, Niš
  - Clinical Centre of Vojvodina, Novi Sad
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Gwangju
  - Department of Oncology, Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Internal Medicine, Seoul
  - Severance Hospital, Seoul
  - St. Mary's Hospital, Seoul
- Switzerland (3):
  - University Hospital Basel, Basel
  - Inselspital, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
- Turkey (Türkiye) (7):
  - Ankara Liv Hospital, Ankara
  - Ankara University Hospital, Ankara
  - Florence Nightingale Hospital, Istanbul
  - Memorial Sisli Hospital, Dept of Hematology, Istanbul
  - Ege University Medical faculty Hospital Internal Medicine Department Adult Hematology Unit, Izmir
  - Izmir Economy University, Medical Point Hospital, Izmir
  - Erciyes University Hospital, Kayseri
- United Kingdom (3):
  - Hammersmith Hospital - Imperial College NHS Healthcare Trust, London
  - University College London (UCL), London
  - The Royal Marsden Hospital, Sutton